CLINICAL TRIAL: NCT00995020
Title: A Study of Two Cone Biopsy Techniques For Women With Cervical Pre-Invasive Disease. LLETZ Cone and SWETZ.
Brief Title: Efficacy Study of Diathermy Cone Biopsy for the Treatment of Cervical Intraepithelial Lesion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, MJCamargo, PHD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 522/99; NCT01733225 (obsolete NCT alias)
Record Dates: First submitted 2009-06-16; First posted 2009-10-14 (Estimated); Results first posted 2012-11-15 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cone biopsy; Conization; Loop electrosurgical excisional procedures; Large Loop Excision of Transformation Zone; Needle Excision of Transformation Zone; Straight Wire Excision of Transformation Zone; Electrosurgery
MeSH Terms: conditions — Uterine Cervical Dysplasia; Hyperthermia | interventions — Conization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SWETZ (Experimental): The intervention administered in this arm is the straight wire excision of the transformation zone, a electrosurgical method to perform a cone biopsy using a 1 cm straight wire of 0.20 mm wire. The activated wire is used in much the same way as a cold knife or laser beam fashioning the surgical specimen to achieve two centimeters cm at cervical canal..
  Interventions: Procedure: Straight Wire Excision of Transformation Zone
- LLETZ cone (Active Comparator): The intervention administered in this arm is the large loop excision of transformation zone as a cone biopsy, performed using a large loop electrode of 2 cm depth, applied to the cervix to achieving two centimeters at cervical canal .
  Interventions: Procedure: Large Loop Excision of Transformation Zone (cone biopsy)

INTERVENTIONS:
Procedure: Straight Wire Excision of Transformation Zone — Straight wire excision of transformation zone is a electrosurgical conization method,which uses a straight wire electrode as a knife to remove the dysplastic epithelium of the cervix.
  Other Names: NETZ - Needle Excision Of Transformation Zone
  Arms: SWETZ
Procedure: Large Loop Excision of Transformation Zone (cone biopsy) — LLETZ cone is a electrosurgical conization method, which is performed with a large loop electrode of 20-25 mm depth. The loop is applied to the cervix outside the lateral margin of TZ and brought slowly to the controlateral TZ margin.
  Other Names: LEEP - Loop Electrosurgical Procedure
  Arms: LLETZ cone

SUMMARY:
The purpose of this trial is to determine whether SWETZ (Straight Wire Excision of Transformation Zone) is a superior alternative to LLETZ cone (Large Loop Excision of Transformation Zone cone biopsy) in the management of pre-invasive endocervical disease.

SWETZ is a new cone biopsy procedure performed with a straight wire electrode and it will be compared to LLETZ cone, which is performed with a large loop electrode.

DETAILED DESCRIPTION:
The treatment of precancerous lesions hinges on the destruction, or more commonly, the excision of the cervical transformation zone . When the transformation zone contains squamous precancer and is completely ectocervical and therefore full visible, excision or destruction is an effective and relatively straightforward therapeutic entity. However in a small proportion of women a cone biopsy is necessary. A cone biopsy often requires the excision of 20-30 mms of endocervical canal.

Interventions.

1. The standard procedure, LLETZ - cone (Large Loop Excision of Transformation Zone cone biopsy), is performed with a large loop electrode of 20-25 mm depth. The activated loop was applied to the cervix outside the lateral margin of transformation zone and brought slowly to the controlateral margin with the objective to acquire 20-25 mm up the canal.
2. The experimental intervention is SWETZ (Straight Wire Excision of Transformation Zone), a method of excision using a 1cm straight disposal of 0.20 wire to remove the endocervical transformation zone or glandular disease. The activated wire was used as a knife, fashioning a cone with desired dimensions.

This technique may be able to excise the endocervical transformation zone with a lower rate of morbidity and incomplete excision rate than LLETZ cone biopsy.

The hypothesis to be tested in this trial is that SWETZ is superior to LLETZ cone in the management of endocervical pre-invasive disease.

ELIGIBILITY:
Inclusion Criteria:

* Incompletely visible transformation zone in women with High grade Squamous Intraepithelial Lesion (HSIL)
* Suspicion of microinvasive carcinoma or occult invasive carcinoma
* Suspicion of glandular disease

Exclusion Criteria:

* Pregnancy
* Coagulation disorders
* Cervicitis were present
* Refusal to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 1999-11; Primary Completion 2004-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: WALTER PRENDIVILLE, PhD, Study Director — British Society of Colposcopy; WALTER PRENDIVILLE, PhD, Study Director — International Federation of Cervical Pathology and Colposcopy
Locations (2):
- Brazil (2):
  - Instituto Fernandes Figueira - Oswaldo Cruz Foundation, Rio de Janeiro, Rio de Janeiro
  - Instituto Fernandes Figueira, Rio de Janeiro, Rio de Janeiro

REFERENCES:
- [Derived] Camargo MJ, Russomano FB, Tristao MA, Huf G, Prendiville W. Large loop versus straight-wire excision of the transformation zone for treatment of cervical intraepithelial neoplasia: a randomised controlled trial of electrosurgical techniques. BJOG. 2015 Mar;122(4):552-7. doi: 10.1111/1471-0528.13200. Epub 2014 Dec 17. PMID 25516462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 1999 and December 2004, patients were assessed for eligibility, the great majority in Rio de Janeiro.
Pre-assignment Details: 127 women were eligible for both arms: 5 refused to participate, 19 did not meet inclusion criteria.
Groups:
- SWETZ - Straight Wire Excision of the Transformation Zone: The experimental intervention was SWETZ (straight wire excision of the transformation zone), which uses a 1cm straight wire electrode to perform a cone. The activated electrode is applied for shaping a cone with the ambition of removing 20-25 mm length of endocervical epithelium.
- LLETZ Cone: Large Loop Excision of Transformation Zone - Cone: The standard procedure, LLETZ - cone (large loop excision of tranformation zone used as cone biopsy), was performed with a large loop electrode of 20-25 mm depth. The activated loop is applied to the cervix outside the lateral margin of TZ (transformation zone) and brought slowly to just outside the controlateral transformation zone margin with the ambition of removing 20-25 mm length of endocervical epithelium.
Period: Overall Study
Arm/Group | SWETZ - Straight Wire Excision of the Transformation Zone | LLETZ Cone: Large Loop Excision of Transformation Zone - Cone
Started | 51 | 52
Completed | 48 (Reasons for not completed: margin analysis not performed specimen fragmentation thermal damage) | 45 (Reasons for not completed: margin analysis not performed specimen fragmentation thermal damage)
Not Completed | 3 | 7
Not completed — margin analysis not performed | 2 | 5
Not completed — specimen fragmentation, thermal damage | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- SWETZ - Straight Wire Excision of the Transformation Zone: The experimental intervention was SWETZ, which uses a 1cm straight wire electrode to perform a cone. The activated electrode is applied for shaping a cone with the ambition of removing 20-25 mm length of endocervical epithelium.
- LLETZ Cone - Loop Excision of TZ Cone Biopsy: The standard procedure, LLETZ - cone, was performed with a large loop electrode of 20-25 mm depth. The activated loop is applied to the cervix outside the lateral margin of TZ and brought slowly to just outside the controlateral TZ margin with the ambition of removing 20-25 mm length of endocervical epithelium.
- Total: Total of all reporting groups
Arm/Group | SWETZ - Straight Wire Excision of the Transformation Zone | LLETZ Cone - Loop Excision of TZ Cone Biopsy | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (9.9) | 45.6 (11.5) | 44.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 46 | 46 | 92
  Ireland | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Endocervical Margin Not Free of Disease.
Description: Primary outcome is the number of participants with incomplete excision of dysplasia at the endocervical excision margin as recognized histologically.
Time Frame: 3 months after the surgery is performed.
Population: All data were analysed bu intention to treat.
Measure: Number; unit: participants
Groups:
- SWETZ: SWETZ (Straight wire excision of the transformation zone), the experimental intervention, is a cone biopsy procedure that uses a 1cm X 0.20mm straight wire to fashion a cone excision,with the ambition of removing 20-25 mm length of endocervical epithelium. Cone biopsy is a surgical procedure which objectives the excision of the pre-invasive disease located at endocervical transformation zone or glandular epithelium of the cervix. This procedure removes the cervical pre-invasive disease for the woman under this condition.
- LLETZ Cone: LLETZ cone,the standard procedure is performed with a large loop electrode of 20-25 mm depth. The activated loop is applied to the cervix outside the lateral margin of TZ and brought slowly to just outside the controlateral TZ margin with the ambition of removing 20-25 mm length of endocervical epithelium.Cone biopsy is a surgical procedure which objectives the excision of the pre-invasive disease located at endocervical transformation zone or glandular epithelium of the cervix. This procedure removes the cervical pre-invasive disease for the woman under this condition.
Arm/Group | SWETZ | LLETZ Cone
Number analyzed (Participants) | 51 | 52
participants | 8 | 10

2. Secondary Outcome: Time Spent to Perform the Procedure
Description: Time was recorded from insertion until removal of the vaginal speculum.
Time Frame: Time spent from randomization to complete the procedure
Measure: Mean (Standard Deviation); unit: minuts
Groups:
- LLETZ - Cone: LLETZ - cone was performed with a large loop electrode of 20-25 mm depth. The activated loop is applied to the cervix outside the lateral margin of TZ and brought slowly to just outside the controlateral TZ margin with the ambition of removing 20-25 mm length of endocervical epithelium.
- SWETZ: SWETZ uses a 1cm straight 0.20mm wire to fashion a similar excision.
Arm/Group | LLETZ - Cone | SWETZ
Number analyzed (Participants) | 52 | 51
minuts | 13.5 (5.3) | 23.2 (8.1)

ADVERSE EVENTS:
Arm/Group | SWETZ - Straight Wire Excision of the Transformation Zone | LLETZ Cone - Loop Excision of TZ Cone Biopsy
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 0/51 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No